CLINICAL TRIAL: NCT01771705
Title: NFAT-Dependent Cytokine Gene Expression for Immune Monitoring in Kidney Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFAT dependent cytokines
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Kidney Transplantation
Keywords: Transplantation; Kidney; calcineurin inhibitor; NFAT; tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose adjust group (NFAT) (Experimental): Within 4 weeks of a 6 month management biopsy, if eligibility is confirmed, NFAT dependent cytokines including IL-2, IFNg, and GMCSF at times C0 and C1.5 will be performed with the residual expression calculated based on the ratio of C1.5/C0 x 100%. If the average residual expression of the 3 cytokines is <20%, the CNI daily dose will be reduced by 15%. If the average residual gene expression of the 3 cytokines is > 60% the CNI daily dose will be increased by 15%.
  Interventions: Other: Dose adjust group (NFAT)
- Standard of care group (No Intervention): A CNI trough level will be obtained. Adjustments of CNI will be based on target trough drug levels as per standard of care.

INTERVENTIONS:
Other: Dose adjust group (NFAT) — If the average residual expression of the 3 cytokines is <20%, the CNI daily dose will be reduced by 15%. If the average residual gene expression of the 3 cytokines is > 60% the CNI daily dose will be increased by 15%.
  Arms: Dose adjust group (NFAT)

SUMMARY:
The purpose of this study is to compare two different ways of monitoring the immune system to determine how to manage the doses of anti-rejection medications.

DETAILED DESCRIPTION:
This is a single center randomized controlled trial investigating the efficacy and safety of adjusting calcineurin inhibitor (CNI) dosing based on Nuclear Factor of Activating T Cells (NFAT)-dependent cytokine gene expression as compared to standard of care adjustments based on trough level. Before any study-related evaluations are performed, the patient must give written informed consent. Once consent is obtained, a patient's eligibility to participate in the study will be assessed within 4 weeks of their 6 month management biopsy. Approximately 40 patients who meet inclusion criteria will be randomized at University of California, San Francisco (UCSF). Eligible patients include any patient maintained on triple therapy with tacrolimus, mycophenolate mofetil ,and prednisone who has had no prior rejection episodes and who has undergone a 6 month management kidney biopsy that shows no evidence of acute cellular rejection or antibody mediated rejection.

ELIGIBILITY:
Inclusion Criteria: Eligible patients include any patient maintained on triple therapy with tacrolimus, mycophenolate mofetil ,and prednisone who has had no prior rejection episodes and who has undergone a 6 month management kidney biopsy that shows no evidence of acute cellular rejection or antibody mediated rejection.

Exclusion Criteria: Any patient not maintained on triple therapy with tacrolimus, mycophenolate mofetil and steroids and/or who had evidence of rejection on 6- month management biopsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05-02 (Actual); Primary Completion 2016-08-13 (Actual); Study Completion 2017-04-17 (Actual)

PRIMARY OUTCOMES:
•Number of adjustments made to tacrolimus regimen at 6 months; •Lack of correlation between NFAT-dependent cytokine expression and tacrolimus trough levels | 6 Months

SECONDARY OUTCOMES:
1 year (18 months post-transplant) biopsy proven acute rejections episodes | 12 Months
1 year (18 months post-transplant) cumulative infectious complications | 12 Months
1 year (18 months post-transplant) GFR | 12 Months
1 year (18 months post-transplant) allograft survival | 12 Months
1 year (18 months post-transplant) patient survival | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, M.D., Principal Investigator — University of California, San Francisco; Allison Webber, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Giese T, Sommerer C, Zeier M, Meuer S. Monitoring immunosuppression with measures of NFAT decreases cancer incidence. Clin Immunol. 2009 Sep;132(3):305-11. doi: 10.1016/j.clim.2009.03.520. Epub 2009 Apr 23. PMID 19398376
- [Result] Giese T, Zeier M, Schemmer P, Uhl W, Schoels M, Dengler T, Buechler M, Meuer S. Monitoring of NFAT-regulated gene expression in the peripheral blood of allograft recipients: a novel perspective toward individually optimized drug doses of cyclosporine A. Transplantation. 2004 Feb 15;77(3):339-44. doi: 10.1097/01.TP.0000109260.00094.01. PMID 14966405
- [Result] Sommerer C, Giese T, Schmidt J, Meuer S, Zeier M. Ciclosporin A tapering monitored by NFAT-regulated gene expression: a new concept of individual immunosuppression. Transplantation. 2008 Jan 15;85(1):15-21. doi: 10.1097/01.tp.0000296824.58884.55. PMID 18192906
- [Result] Sommerer C, Zeier M, Meuer S, Giese T. Individualized monitoring of nuclear factor of activated T cells-regulated gene expression in FK506-treated kidney transplant recipients. Transplantation. 2010 Jun 15;89(11):1417-23. doi: 10.1097/TP.0b013e3181dc13b6. PMID 20463649
- [Result] Hartmann B, Schmid G, Graeb C, Bruns CJ, Fischereder M, Jauch KW, Heeschen C, Guba M. Biochemical monitoring of mTOR inhibitor-based immunosuppression following kidney transplantation: a novel approach for tailored immunosuppressive therapy. Kidney Int. 2005 Dec;68(6):2593-8. doi: 10.1111/j.1523-1755.2005.00731.x. PMID 16316335
- [Result] Leogrande D, Teutonico A, Ranieri E, Saldarelli M, Gesualdo L, Schena FP, Di Paolo S. Monitoring biological action of rapamycin in renal transplantation. Am J Kidney Dis. 2007 Aug;50(2):314-25. doi: 10.1053/j.ajkd.2007.05.002. PMID 17660033
- [Result] Belouski SS, Wilkinson J, Thomas J, Kelley K, Wang SW, Suggs S, Ferbas J. Utility of lyophilized PMA and ionomycin to stimulate lymphocytes in whole blood for immunological assays. Cytometry B Clin Cytom. 2010 Jan;78(1):59-64. doi: 10.1002/cyto.b.20492. PMID 19777549